CLINICAL TRIAL: NCT00516581
Title: Occurrence of Pneumocystis Pneumonia in HIV-Infected Patients and the Interference of the Highly Active Antiretroviral Therapy
Brief Title: Occurrence of Pneumocystis Pneumonia in HIV-Infected Patients and the Interference of the HAART
Status: Completed | Type: Observational
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Responsible Party: Sergio Muller, Faculdade de Medicina de Botucatu - Unesp
Other Study IDs: upeclin/HC/FMB-Unesp-13; PCP UnespFMB 2003
Record Dates: First submitted 2007-08-14; First posted 2007-08-15 (Estimated); Last update posted 2008-09-05 (Estimated); Status verified 2008-09

CONDITIONS: HIV
Keywords: Pneumocystis Pneumonia; Acquired Immune Deficiency Syndrome; Highly Active Antiretroviral Therapy; Treatment Experienced; Treatment Naive
MeSH Terms: conditions — Pneumonia, Pneumocystis; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- no HAART: Patients that no received HAART
- with HAART: Patients that received HAART

SUMMARY:
From the beginning of the AIDS epidemic, pulmonary pneumocystosis (PCP) has been distinguished as one of the most frequent opportunistic diseases with high morbid-mortality. As from 1996, the advent of the highly active antiretroviral therapy (HAART) has changed the characteristics of such epidemic by reducing its related diseases and, as a result, AIDS-related mortality. With the purpose to estimate PCP occurrence and HAART interference, 376 HIV-infected or AIDS patients were studied from January 1992 to December 2002.

DETAILED DESCRIPTION:
From the beginning of the AIDS epidemic, pneumocystis pneumonia (PCP) has been distinguished as one of the most frequent opportunistic diseases with high morbid-mortality. As from 1996, the advent of the highly active antiretroviral therapy (HAART) has changed the characteristics of such epidemic by reducing its related diseases and, as a result, AIDS-related mortality. With the purpose to estimate PCP occurrence and HAART interference, 376 HIV-infected or AIDS patients were studied from January 1992 to December 2002. Among them, 58 (15.5%) PCP cases were found. There was a higher occurrence of PCP in the group of patients in which HAART was not used, with 40 (69.0%) of the episodes. As regards the studied period, a tendency to a linear reduction in annual PCP incidence was observed. The mean of T CD4+ lymphocytes in the patients with PCP (117 cells/mm3) was significantly lower when compared to that of the other individuals (325 cells/mm3). Therefore, this study suggests a temporal reduction in PCP occurrence related to HAART use with higher T CD4+ lymphocyte counts. Nevertheless, this opportunistic infection still shows significant incidence in AIDS patients.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection

Exclusion Criteria:

* No HIV infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 376 HIV-infected or AIDS patients were studied from January 1992 to December 2002
Sampling Method: Probability Sample
Enrollment: 376 (Actual)
Dates: Start 2003-02; Study Completion 2005-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre N Barbosa, MD, MSc, Principal Investigator — UPECLIN HC FM Botucatu Unesp
Locations (1):
- Faculdade de Medicina de Botucatu - Unesp, Botucatu, São Paulo, Brazil